CLINICAL TRIAL: NCT04566302
Title: Pilot Study of Imaging Human Skin With High-Speed Spectrally Encoded Confocal Microscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Principal Investigator - MD, PhD, FACC, FCAP, FNAI, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2019P001237
Record Dates: First submitted 2020-08-11; First posted 2020-09-28 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Pigmented Lesions; Pigmented Skin Lesion; Pigmented Moles; Skin Lesion
Keywords: SECM; Spectrally Encoded Confocal Microscopy; RCM; Reflectance Confocal Microscopy
MeSH Terms: conditions — Nevus, Pigmented

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- SECM Skin Imaging (Experimental): The SECM skin imaging procedure will be very similar to that by the FDA approved RCM devices. First, the skin lesion (such as a mole) will be identified on a forearm of the subject. The lesion will be imaged first with a dermatoscope, and then with the SECM device. A dermatoscope is a hand-held device used for the visual observation of the epidermis. It is a superior surface contact microscope used to examine skin lesions.
  Interventions: Device: SECM Skin Imaging

INTERVENTIONS:
Device: SECM Skin Imaging — Consented Participants will be asked to allow their forearm to be imaged by the dermatoscope on the same skin/lesions as a control comparison. We will be trying to image pigmented skin/lesions present on the forearm. This will be followed by imaging using the SECM Skin imaging device

SUMMARY:
The aim of this study is to evaluate the imaging performance of Spectrally Encoded Confocal Microscopy (SECM) for imaging human skin and skin diseases.

DETAILED DESCRIPTION:
SECM provides an order of magnitude faster imaging speed than conventional confocal microscopy devices. The investigators have previously utilized the SECM technology for imaging large area of human esophagus in vivo. They have also developed endoscopic capsule devices which have been used to safely image over 60 human subjects, healthy volunteers and subjects with eosinophilic esophagitis, using SECM technology, rapidly.

When used for skin imaging, SECM can provide real-time three-dimensional confocal imaging and significantly reduce the imaging time. While SECM has been successfully used for imaging human esophagus in vivo, its utility in skin imaging needs to be tested in a new pilot study. The investigators will be taking images with a dermatoscope as well. This will the control to compare the experimental images to, as the dermatoscope is the standard of care diagnostic tool for dermatologists.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* 18 years of age or older
* Capable of giving informed consent
* Pigmented lesions (such as moles) present on the forearm

Exclusion Criteria:

* Unable to provide consent
* Open cuts/sores on the skin, skin infection, or any contagious skin condition
* Pregnant women (according to subject)
* Employees under the direct supervision of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, M.D, PhD., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SECM Skin Imaging
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SECM Skin Imaging
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 36.875 [23 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Quality Skin Images Obtained From SECM Device
Time Frame: Approximate 30 minute study
Population: 15 participants were imaged with both SECM device and dermatoscope.
Measure: Count of Participants; unit: Participants
Groups:
- SECM Skin Imaging: The SECM skin imaging procedure will be very similar to that by the FDA approved RCM devices. First, the skin lesion (such as a mole) will be identified on a forearm of the participant. The lesion will be imaged first with a dermatoscope, and then with the SECM device. A dermatoscope is a hand-held device used for the visual observation of the epidermis. It is a superior surface contact microscope used to examine skin lesions.
Arm/Group | SECM Skin Imaging
Number analyzed (Participants) | 15
Participants | 15

ADVERSE EVENTS:
Time Frame: Imaging data is collected during the procedure (up to 30 minutes).
Description: Other Adverse Event
Arm/Group | SECM Skin Imaging
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SECM Skin Imaging (N=16)
Mild, self resolving skin discomfort prior to imaging (Skin and subcutaneous tissue disorders) | 1 (1) — Mild skin discomfort prior to imaging, not affecting subject safety, resolved without intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT04566302/Prot_SAP_000.pdf